CLINICAL TRIAL: NCT07322419
Title: Echocardiographic Evaluation of Cardiac Output During Cesarean Delivery Under Spinal Anesthesia Using Norepinephrine Versus Ephedrine: A Randomized Controlled Trial
Brief Title: Hemodynamics During Cesarean Delivery Under Spinal Anesthesia With Norepinephrine Versus Ephedrine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD.25.04.982
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery; Spinal Anesthesia for Cesarean Section
Keywords: Cesarean delivery; Spinal anesthesia; Echocardiography; Hemodynamics
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine; Fentanyl; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine (Experimental)
  Interventions: Procedure: Spinal Anesthesia with Bupivacaine and Fentanyl; Drug: Crystalloid Coload 1000 mL; Procedure: Cesarean Delivery; Radiation: Transthoracic Echocardiography; Drug: Intravenous Norepinephrine Bolus
- Ephedrine (Active Comparator)
  Interventions: Procedure: Spinal Anesthesia with Bupivacaine and Fentanyl; Drug: Crystalloid Coload 1000 mL; Procedure: Cesarean Delivery; Radiation: Transthoracic Echocardiography; Drug: Intravenous Ephedrine Bolus

INTERVENTIONS:
Procedure: Spinal Anesthesia with Bupivacaine and Fentanyl — Spinal anesthesia using 2.5 mL of 0.5% hyperbaric bupivacaine (12.5 mg) and 15 mcg of fentanyl at the L4-L5 or L3-L4 interspace
Drug: Crystalloid Coload 1000 mL — Ringer acetate 1000 mL will be administered over 10 minutes starting immediately after intrathecal injection
Procedure: Cesarean Delivery — Lower segment cesarean section using the Pfannenstiel incision and uterine exteriorization
Radiation: Transthoracic Echocardiography — Measurement of cardiac output in supine position with left lateral tilt at baseline, at 1 and 10 minutes after intrathecal injection, and immediately after delivery
Drug: Intravenous Norepinephrine Bolus — Prophylactic IV norepinephrine bolus of 6 mcg will be administered immediately after intrathecal injection, followed by rescue IV norepinephrine boluses of 3, 6, and 9 mcg when systolic blood pressure decreases below 90%, 80%, and 70% of baseline value, respectively
  Arms: Norepinephrine
Drug: Intravenous Ephedrine Bolus — Prophylactic IV ephedrine bolus of 6 mg will be administered immediately after intrathecal injection, followed by rescue IV ephedrine boluses of 3, 6, and 9 mg when systolic blood pressure decreases below 90%, 80%, and 70% of baseline value, respectively
  Arms: Ephedrine

SUMMARY:
Echocardiography will be used to measure cardiac output and calculate other important hemodynamic variables in healthy patients with full-term singleton pregnancy during cesarean delivery under conventional spinal anesthesia using 2 different vasopressor drugs: norepinephrine in 1 group versus ephedrine in another group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II.
* Singleton, full term pregnancy.
* Scheduled cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* Height <150 or >180 cm.
* Weight <60 or >110 kg.
* Body mass index (BMI) <18.5 or ≥35 kg/m².
* Women presenting in labor.
* Any contraindication to spinal anesthesia: increased intracranial pressure, coagulopathy, or local skin infection.
* Chronic or pregnancy-induced hypertension.
* Baseline systolic blood pressure >140 mm Hg.
* Hemoglobin <10 g/dl.
* Diabetes mellitus, cardiovascular, cerebrovascular, or renal disease.
* Polyhydramnios or known significant fetal abnormalities.
* Current administration of vasoactive drugs such as: beta blockers, salbutamol, or thyroxin.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between the 2 groups in cardiac output at 10 minutes after intrathecal injection | From the start of spinal anesthesia until delivery

SECONDARY OUTCOMES:
Differences between the 2 groups in cardiac output at 1 minute after intrathecal injection and after delivery | From the start of spinal anesthesia until delivery
Differences between the 2 groups in stroke volume at 1 and 10 minutes after intrathecal injection, and after delivery | From the start of spinal anesthesia until delivery
Differences between the 2 groups in heart rate at 1 and 10 minutes after intrathecal injection, and after delivery | From the start of spinal anesthesia until delivery
Differences between the 2 groups in mean arterial pressure at 1 and 10 minutes after intrathecal injection, and after delivery | From the start of spinal anesthesia until delivery
Differences between the 2 groups in systemic vascular resistance at 1 and10 minutes after intrathecal injection, and after delivery | From the start of spinal anesthesia until delivery
Number of patients receiving rescue vasopressor | From the start of spinal anesthesia until delivery
  Systolic blood pressure <90% of baseline value
Incidence of hypotension | From the start of spinal anesthesia until delivery
  Systolic blood pressure <80% of baseline value
Incidence of severe hypotension | From the start of spinal anesthesia until delivery
  Systolic blood pressure <70% of baseline value
Incidence of bradycardia | From the start of spinal anesthesia until delivery
  Heart rate <50 beats/min
Incidence of nausea and/or vomiting | From the start of spinal anesthesia until delivery
Total vasopressor dose | From the start of spinal anesthesia until delivery
Neonatal Apgar score at 1 and 5 minutes after delivery | 1 and 5 minutes after delivery
  Scale from 0 to 10. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Surgical Critical Care, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be provided to the Publishing journal if requested